CLINICAL TRIAL: NCT01777178
Title: Intradialytic Acid-base Changes and Organic Anion Production With Standard Versus Low Bicarbonate Hemodialysis
Brief Title: Comparison of Standard Versus Low Bicarbonate Hemodialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Matthew Abramowitz, Assistant Professor, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-684
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2013-06

CONDITIONS: Chronic Kidney Disease; Metabolic Acidosis
Keywords: bicarbonate; dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low bicarbonate dialysis (Experimental)
  Interventions: Other: Low bicarbonate dialysis

INTERVENTIONS:
Other: Low bicarbonate dialysis

SUMMARY:
This study will compare acid-base changes during hemodialysis treatments with a standard dialysis bath versus a lower bicarbonate dialysis bath, and aims to define the factors that limit equilibration of the bicarbonate concentration in a patient's blood with that in the dialysate.

ELIGIBILITY:
Inclusion Criteria:

* Receiving chronic thrice-weekly conventional hemodialysis for at least 3 months
* Age > 18 years

Exclusion Criteria:

* Use of oral alkali within the previous month
* Hospitalization within the previous month
* Inability to provide written informed consent
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in beta-hydroxybutyrate clearance | 1-2 weeks
  Comparison between 2 hemodialysis treatments with different bicarbonate dialysis concentrations
Change in lactate clearance | 1-2 weeks
  Comparison between 2 hemodialysis treatments with different bicarbonate dialysis concentrations
Post-dialysis pH | 1-2 weeks
Post-dialysis bicarbonate | 1-2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew K Abramowitz, MD, MS, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center/Jack D. Weiler Hospital, The Bronx, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2013-01-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT01777178/ICF_000.pdf